CLINICAL TRIAL: NCT02467088
Title: An Observational Study on the Efficacy of Individualised Homoeopathic Treatment on Premenstrual Syndrome in Indian Females
Brief Title: An Observational Study on the Efficacy of Individualised Homoeopathic Treatment on Premenstrual Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr J. Pellow, University of Johannesburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MaseehaBulbulia200700939
Record Dates: First submitted 2015-05-14; First posted 2015-06-09 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; Individualised homoeopathic treatment; Indian females
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Individualised Homoeopathic Remedy (Experimental): Each participant will receive an individualised homoeopathic remedy, in a vehicle of sucrose pillules, according to the symptoms of their PMS. Although different individualised remedies may be dispensed, each remedy will be homoeopathic. Each individualised homoeopathic remedy will have an individualised dosage, frequency and duration based on the laws of individualised homoeopathic prescribing as outlined by De Schepper.
  Interventions: Other: Individualised Homeopathic Remedy

INTERVENTIONS:
Other: Individualised Homeopathic Remedy — Each participant will receive an individualised homoeopathic remedy prescribed according to the individualised symptoms of their PMS.

SUMMARY:
Premenstrual Syndrome (PMS) is a group of physical, mental and behavioural symptoms that occur cyclically through the luteal phase of the menstrual cycle and resolve within three days of the onset of menstruation. Many women are affected by the physical and psychological symptoms of PMS. The symptoms of PMS can change behaviour and wellbeing of women which has an impact on families, social life and work. Research has shown that women with PMS reported additional days missed at work compared to women that do not suffer with PMS. A study done by Brohi et al. (2011) showed that PMS is a common problem that occurs in 81.25% of women and has an adverse impact on a woman's quality of life. Conventional treatment is limited, not always effective and is associated with many side effects. Research using individualised homeopathic treatment, known as the homeopathic similimum, in PMS has shown to be well tolerated as well as have a positive impact on the symptoms of PMS although further research is warranted in this regard. There have not been any studies done on homeopathic treatment in Indian females in South Africa.

The aim of this study is to determine the effect of individualised homeopathic treatment on females of Indian origin who are suffering with symptoms of PMS, using observational studies.

DETAILED DESCRIPTION:
This study will be a 12 week observational study of an embedded mixed method design and will be conducted over 12 weeks, consisting of four consultations 4 weeks apart, at the Homeopathic Health Centre, University of Johannesburg Doornfontein Campus. Ten South African Indian females, between 18-40 years of age, who experience PMS symptoms will be recruited through the placement of advertisements placed at health stores, homoeopathic/medical practices and on the University campus (with the relevant permission granted).

Each participant must meet the criteria of the selection questionaire. In the first consultation, the researcher will explain the study to the participant. The participant will then be requested to sign the Participant Information and Consent Form. A full case history will be taken using a standard homeopathic case taking form. Each participant will be given a PMS chart to score their symptoms every day for the following 4 weeks in order to establish the baseline of each participant's premenstrual symptoms. No treatment will be prescribed in this period.

Participants will be reminded of their appointments via email and text message before every follow up consultation. Each follow-up consultation will consist of a homoeopathic case taking, relevant physical examination and the collection of the PMS-chart which was completed over the previous 4 weeks by the participant.

After each follow-up consultation, the researcher will establish the participant's individualised homoeopathic remedy according to the principles of classical homoeopathy by using the Complete Repertory 2014 provided in Mercurius® repertory software and the standard Materia Medica, with the guidance of the supervisor or co-supervisor. The potency and dosage of each remedy will be determined in accordance with the principles of individualised homoeopathic prescribing as described by De Schepper. The selected remedy will then be dispensed to the participant. No remedy will be dispensed at week 12. The participant will return a completed PMS-chart, completed over a 4 week period, to the researcher at weeks 4, 8 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Females between ages of 18 and 40 years who experience PMS on a monthly basis;
* females who experience an increase in at least one of the following mental and physical symptoms at least fourteen days before their menses begin, in each of the three preceding menstrual cycles: Mental symptoms: irritability, depression or anxiety Physical symptoms: breast tenderness or swelling, abdominal bloating, headaches, swelling of extremities or food cravings; and
* females who have an amelioration of the above symptoms within three days of the onset of menses and symptoms should not reoccur until at least day thirteen of the cycle.

Exclusion Criteria:

* Irregular menstrual cycles;
* lactating females;
* prediagnosed anxiety and depression;
* use of sex hormones except the oral contraceptive (must have been used for a minimum of 3 months) or concomitant psychotherapies and alternate therapies for PMS
* pregnant females

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
PMS symptoms severity on PMS chart | 12 weeks
  The PMS chart will be completed every day for 12 weeks, recording the participant's symptoms based on the most characteristic PMS symptoms and has been used in previous PMS studies. The evaluation of symptoms is subjective and is based on a 5 point scale: 0 - "no symptom", 1- "very mild", 2 - "mild", 3 - "severe", 4 - "extremely severe".

SECONDARY OUTCOMES:
Case notes on patient symptoms and wellbeing | 12 weeks
  Qualitative data will be collected by the researcher from the participant at weeks 0, 4, 8 and 12 using case notes.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Patel, MTech.Hom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No